CLINICAL TRIAL: NCT01943162
Title: Enhanced Cognitive Rehabilitation to Treat Comorbid TBI and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego Veterans Healthcare System (U.S. Federal Agency)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy Jak, Staff Neuropsychologist, San Diego Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-11-1-0641
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: PTSD With a History of Mild to Moderate TBI
MeSH Terms: interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART-CPT (Experimental): CPT with additional elements of cognitive rehabilitation
  Interventions: Behavioral: CPT
- CPT (Active Comparator): Standard Cognitive Processing Therapy
  Interventions: Behavioral: CPT

INTERVENTIONS:
Behavioral: CPT

SUMMARY:
This study will test a modification of Cognitive Processing Therapy (CPT) for Post-Traumatic Stress Disorder, (PTSD) in which CPT is augmented with compensatory cognitive rehabilitation principles from the Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) intervention to create a hybrid treatment, SMART-CPT. This study investigates the efficacy of SMART-CPT in improving PTSD and post-concussive symptoms, cognition, quality of life, and treatment compliance in those with a history of mild to moderate TBI and persistent cognitive complaints.

ELIGIBILITY:
Inclusion Criteria:

1) OEF/OIF veteran; 2) Current diagnosis of PTSD; 3) History of mild-to-moderate TBI; 4) Subjective cognitive complaints; 5) No anticipated/pending medication changes; 6) Written informed consent to participate in the study. -

Exclusion Criteria:1) Active substance dependence, 2) Suicidal intent or attempt within the previous month; 3) Current psychotic disorder; 4) Dementia; 5) Non-English speaking; 6) Participation in other intervention studies.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2012-08; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist | change from baseline PTSD Checklist at 12 weeks (post-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Jak, Ph.D., Principal Investigator — VA San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Derived] Crocker LD, Sullan MJ, Jurick SM, Thomas KR, Davey DK, Hoffman SN, Twamley EW, Jak AJ. Baseline executive functioning moderates treatment-related changes in quality of life in veterans with posttraumatic stress disorder and comorbid traumatic brain injury. J Trauma Stress. 2023 Feb;36(1):94-105. doi: 10.1002/jts.22883. Epub 2022 Oct 6. PMID 36204974